CLINICAL TRIAL: NCT04243057
Title: Diagnosis, Treatment Status and Prognosis of Cholangiocarcinoma in China: a Multicenter, Two-way, Non-intervention Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Dong Jiahong, Executive President of Beijing Tsinghua Changgung Hospital, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: RWS-BTCH-001
Record Dates: First submitted 2020-01-24; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, two-way, non-intervention study. the main purpose: Understand the current status of diagnosis and treatment of cholangiocarcinoma patients in China and observe the effect of different treatment options on patient recurrence and long-term survival

Secondary purpose:

1. Exploring the actual clinical treatment situation and its compliance with the existing diagnosis and treatment of bile duct cancer
2. Exploring the establishment of clinical research standard fields and standards for diagnosis and treatment of bile duct cancer

ELIGIBILITY:
Inclusion Criteria:

1. above the age of 18 years old, male or female
2. clinical diagnosis of patients with cholangiocarcinoma
3. Child-Pugh classification of A, B
4. Eastern Cooperative Oncology Group scoring system (ECOG) score of 0-2 points

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from 21 hospitals limit:5000
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
RFSR | 3 years
  RFSR-Recurrence Free Survival Rate

SECONDARY OUTCOMES:
OS | 3 years
  OS-Overall Survival
RFS | 3 years
  RFS-Recurrence Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No